CLINICAL TRIAL: NCT05575622
Title: Clinical Study for Combined Analysis of CTC and Exosomes on Predicting the Efficacy of Immunotherapy in Patients With Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20221002
Record Dates: First submitted 2022-10-03; First posted 2022-10-12 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with hepatocellular carcinoma receiving immunotherapy
  Interventions: Device: CTC PD-L1, exosomal PD-L1, and exosomal LAG-3 detection

INTERVENTIONS:
Device: CTC PD-L1, exosomal PD-L1, and exosomal LAG-3 detection — Collect peripheral blood sample of 200 HCC patients at treatment baseline, every time point response till disease progression.Blood samples will be transferred to central lab to detect CTC PD-L1, exosomal PD-L1, and exosomal LAG-3 by microfluidic chip.Tumor response evaluation will be performed after two cycles of therapy by CT/MRI based on RECIST.Clinical data, including tumor stage,metastatic organ ,regimen, objective response, progression free survival, overall survival, etc, will be collected according to study protocol.

SUMMARY:
This project intends to perform CTC PD-L1 imaging, exosomal PD-L1 protein detection, and exosomal LAG-3 protein detection, so as to resolve the functional marker profiles of immunotherapy in the peripheral blood of HCC patients and comprehensively present the responsiveness of patients to immunotherapy.

DETAILED DESCRIPTION:
Liquid biopsy methods such as PD-L1 of CTC, number of peripheral immune cells and their subtypes, and exosomal PD-L1 provide a dynamic monitoring strategy for immunotherapy evaluation. Monitoring CTC and immune-related functional markers in peripheral blood can dynamically reflect the multi-dimensional characteristics of tumor microenvironment, comprehensively represent the response of patients to immunotherapy, and provide a new strategy of companion diagnostics for immunotherapy in HCC. This project intends to perform CTC PD-L1 imaging, exosomal PD-L1 protein detection, and exosomal LAG-3 protein detection, so as to resolve the functional marker profiles of immunotherapy in the peripheral blood of HCC patients and comprehensively present the responsiveness of patients to immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* having signed informed consent
* clinically or pathologically confirmed hepatocellular carcinoma;
* liver tumor load not exceeding 50% of liver volume;
* expected survival ≥ 12 weeks;
* vital organ function meeting enrollment criteria; and (6) no need for pregnancy.

Exclusion Criteria:

* Patients who have been diagnosed with malignant tumors of other systems or organs;
* Patients with hematologic disorders and extreme physical failure;
* Patients with immune deficiencies or organ transplants;
* Other conditions deemed by the investigator to be inappropriate for participation in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in this study were enrolled by the Clinical Trial Centerin Zhongnan Hospital.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
CTC-PD-L1, exosomal PD-L1, and exosomal LAG-3 | Treatment baseline; Up to 2 months from the initial treatment; From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months

CONTACTS AND LOCATIONS:
Overall Officials: Fubing Wang, Doctor, Study Director — Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China